CLINICAL TRIAL: NCT00097396
Title: A Phase 1, Open-Label, Dose-Escalating Study to Evaluate the Safety, Tolerability and Immunogenicity of the Recombinant Plague Vaccine rF1V in Healthy Volunteers
Brief Title: Safety, Tolerability & Immunogenicity of the Recombinant Plague Vaccine rF1V
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Responsible Party: Chief Medical Officer, DynPort Vaccine Company, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rF1V-01
Record Dates: First submitted 2004-11-23; First posted 2004-11-24 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Pneumonic Plague; Preventive Therapy
Keywords: plague; recombinant plague vaccine; vaccine; plague vaccine; Protection against pneumonic plague
MeSH Terms: conditions — Plague

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: rF1V vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a two-dose schedule of the recombinant plague vaccine rF1V in healthy volunteers when given as an intramuscular (IM) injection at four ascending dose-levels. The purpose of the Cohort 4 Extension is to evaluate the safety and tolerability of a third intramuscular (IM) dose of 160 ug rF1V in healthy volunteers who have previously been vaccinated with the same concentration of rF1V vaccine.

DETAILED DESCRIPTION:
The Phase 1 clinical trial is designed as an open-label, single-center, dose-escalation study to evaluate the safety, tolerability, and immunogenicity of a two-dose regimen of rF1V in healthy volunteers at four dose-levels (20 ug, 40 ug, 80 ug and 160 ug rF1V) in four sequential cohorts. The protocol was amended 26 January 2006 to recruit volunteers from Cohort 4 to participate in an Extension. Cohort 4 Extension volunteers will receive a third vaccination at day E-0. Day E-0 (-1) should not exceed Day 240 of the Phase 1 study.

ELIGIBILITY:
Inclusion Criteria:

* The volunteer is male or female and 18 to 40 years of age (inclusive) at the time of the first dose of investigational product
* Good health as determined by screening medical history and physical examination
* The volunteer has the following laboratory parameters within normal range: total WBC, Hemoglobin, platelets, LFT (AST, ALT, ALP, Bilirubin) and/or ≤ 1+ proteinuria. Other laboratory parameters must be within 10 % of the upper or lower limits of the normal range of the University of Kentucky clinical laboratory and not clinically significant as assessed by the Investigator and/or Sponsor Medical Monitor.
* The volunteer has a normal electrocardiogram (ECG). However, if a potential volunteer is reported to have a benign ECG abnormality (e.g., sinus bradycardia) the results may be discussed with the Sponsor Medical Monitor and Covalent Medical Monitor. With the agreement of the Investigator, Covalent Medical Monitor and Sponsor Medical Monitor and documentation of the consultation in the volunteer's study record the Investigator may include the volunteer in the study.
* The volunteer is willing to have his or her blood samples stored for future plague research studies.
* The volunteer has signed the Informed Consent Form, successfully completed (at least 90 % correct) the Test of Understanding, and has signed the HIPAA authorization form.
* The volunteer agrees not to donate blood for at least 30 days following vaccination.
* The volunteer is willing to comply with the requirements of the protocol through the post-vaccination Day 180 (± 7 days) visit.
* Female volunteers must be of non-childbearing potential (i.e., surgically sterilized or postmenopausal), or must not be pregnant (as indicated by a negative serum pregnancy test within 24 hours prior to rF1V administration) or nursing, and must use two types of an acceptable form of FDA-approved contraception (barrier method, Depo-Provera, Norplant, Ortho Evra (birth control patch), oral contraceptives) through 30 days after the second (final) vaccination of rF1V (i.e. Day 58). If abstinent, two forms of birth control are not required

Inclusion Criteria (Cohort 4 Extension)

* The volunteer must be an active participant enrolled in Phase 1 rF1V-01 protocol - Cohort 4 (160 ug) completing day 180 procedures as defined in rF1V-01 protocol
* Have good health as determined by screening medical history and physical examination
* Have a blood potassim level of no less than 3.6 mEq/mL and have no clinically significant abnormalities on other laboratory safety tests from the study Day 180 assessments
* The volunteer has signed the informed consent form for Cohort 4 Extension
* The volunteers agrees not to donate blood for at least 30 days following vaccination
* The volunteer is willing to comply with the requirements of the protocol from the day of vaccination Study Day E-0 (-1) through Study Day E-180 (+/- 14 days)final visit
* Female volunteers must be of non-childbearing potential (i.e., surgically sterilized or postmenopausal), or must not be pregnant (as indicated by a negative blood pregnancy test within one day prior to rF1V administration) or nursing, and must use two types of an acceptable form of FDA-approved contraception (barrier method, Depo-Provera, Norplant, Ortho Evra (birth control patch), oral contraceptives) through 30 days after vaccination with rF1V (i.e. Study Day E-30). If abstinent, two forms of birth control are not required

Exclusion Criteria:

* Have a history of plague disease or have received any plague vaccine.
* Have active tuberculosis or other systemic infectious process by review of systems and physical examination.
* Have a history of allergy to kanamycin or aminoglycosides.
* Positive for human immunodeficiency virus (HIV); hepatitis C virus (HCV) or hepatitis B surface antigen (HbsAg)
* Have a history of immunodeficiency, chronic illness requiring continuous or frequent medical intervention, acute/chronic untreated conditions, autoimmune disease, or use of immunosuppressive medications.
* The volunteer has chronic, severe or recurrent joint pain or arthritis of any etiology.
* The volunteer has a positive result on a urine drug screen that tests for common substances of abuse such as amphetamines, barbiturates, benzodiazepines, cocaine, opiates, and cannabinoids. (If positive on screen, confirmatory testing shall be performed where applicable).
* The volunteer has previous diagnosis of any serious psychiatric disorder. For this purpose, serious psychiatric disorder is defined as illness requiring hospitalization within the previous 12 months; routine administration of more than one medication to control anxiety, mood or sleep disorder; or history of suicide attempt.
* The volunteer has received any blood products or immune globulin in the previous six months.
* The volunteer has donated blood within the past 56 days.
* The volunteer received any investigational drug therapy within 30 days before the first dose of rF1V or intends to receive any other investigational drug therapy before the post-vaccination Day 180 (± 7 days) visit.
* The volunteer has a clinically significant abnormality on the ECG.
* The volunteer has a body mass index 40 kg/m2 or is greater than or equal to 100 lbs over the ideal body weight.
* The volunteer has an acute illness, evidence of significant active infection, or evidence of systemic disease at time of enrollment that in the opinion of the Investigator would place the volunteer at an unacceptable risk for injury.
* Have temperature greater than or equal to 100º F on the day of scheduled 1st vaccination.
* Have personal history of multiple sclerosis, since immune system stimulation may exacerbate this disorder.
* Have occupational or other responsibilities that would prevent completion of participation in the study.
* Licensed vaccines are not exclusionary but should be given at least 2 weeks before or after immunization (if live vaccine: 60 days before or after immunization) to avoid potential confusion of adverse reactions.
* Screening laboratory values for total WBC, Hemoglobin, platelets, LFT (AST, ALT, ALP, Bilirubin) are not within normal range and/or more than 1+ proteinuria.
* Have a history of anaphylaxis or other serious adverse reactions to vaccines.
* The female volunteer is pregnant (must have a negative serum pregnancy test within 24 hours prior to each dose of rF1V), lactating or unwilling to use two types of an acceptable form of FDA-approved contraception through 30 days after the second (final) dose of rF1V (i.e. Day 58)
* Are receiving ongoing chemotherapy with immunosuppressive agents such as systemic corticosteroids within 3 months prior to or during the study.
* A total steroid dose of 2mg/kg or 20mg/day within 3 months (ACIP recommendation) and "Burst" therapy within 2 weeks prior to vaccination is permitted. Inhaled and topical steroids are permitted.
* Veterans with prior record of receiving any plague vaccine

Exclusion Criteria (Cohort 4 Extension)

* Not currently enrolled in Cohort 4 of the rF1V-01 protocol
* The volunteer received any investigational drug therapy (other than that received in the rF1V-01 study) within 30 days before vaccination with rF1V or intends to receive any other investigational drug therapy before the post-vaccination Study Day E-180 (+/- 14 days) visit
* Blood potassium level is below 3.6 mEq/L on Study Day 180 safety laboratory test or other safety laboratory values from rF1V-01 Study Day 180 (+/- 7 days) or later have clinically significant abnormalities
* The female volunteer is pregnant (must have a negative blood pregnancy test within one day prior to receipt of rF1V), lactating or unwilling to use two types of an acceptable for of FDA-approved contraception through 30 days after vaccination with rF1V (i.e., Study Day E-30)
* Have received a total prednisone-equivalent corticosteroid dose of greater than or equal to 2mg/kg or 20mg/day within 3 months (ACIP recommendation) or "Burst" therapy within 2 weeks prior to vaccination. Inhaled and topical steroids are permitted
* Have previously received any plague vaccine other than two doses of rF1V (160 ug)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2004-11; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of a two-dose schedule of the recombinant plague vaccine rF1V in healthy volunteers when given as an IM injection at four ascending dose-levels.

SECONDARY OUTCOMES:
To evaluate immunogenicity of a two-dose schedule of rF1V vaccine when given as an IM injection at four ascending dose-levels
To collect and store serum samples for future immunogenicity assays (e.g. ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Greenberg, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- See also: sponsor website — http://www.dynport.com